CLINICAL TRIAL: NCT04209621
Title: Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to unexpected sudden death on study.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Clare Sun, M.D., Staff Clinician, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200016; 20-H-0016
Record Dates: First submitted 2019-12-21; First posted 2019-12-24 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Small Lymphocytic Leukemia (SLL); Chronic Lymphocytic Leukemia (CLL)
Keywords: P13K Inhibitor; PLCG2 Mutations; BTK Mutations; Myeloid Cells and Myeloid Derived Suppressor Cells (MDSCs); T and Leukemic B Cells Aggregate
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — duvelisib; ibrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (Other): Duvelisib with ibrutinib will be administered for the first six 28-day (± 7) cycles followed by duvelisib alone until disease progression or intolerance. Duvelisib is an orally administered at 15 mg twice a day (dose level 1) or 25 mg twice day (dose level 2). Subjects will continue the same dose of ibrutinib prior to study enrollment for the first six 28-day cycles. Ibrutinib is an orally administered and provided as 140 mg white opaque capsules or tablets in 4 strengths: 140 mg, 280 mg, 420 mg, and 560 mg.
  Interventions: Drug: Duvelisib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Duvelisib — twice daily as tolerated until disease progression
  Other Names: Copiktra
Drug: Ibrutinib — daily for the first six 28-day cycles
  Other Names: Imbruvica

SUMMARY:
Background:

Chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) are cancers often treated with the drug ibrutinib. For some people, ibrutinib stops working. Researchers want to see if adding another drug can help.

Objective:

To test how people with ibrutinib-resistant CLL respond to duvelisib.

Eligibility:

People ages 18 and older with CLL or SLL that is no longer responding to ibrutinib or has developed mutations that could stop it from working

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Heart tests
* Blood and urine tests
* CT scan. For this, participants will have a dye injected into a vein. They will lie in a machine that takes pictures of the body.
* Bone marrow biopsy. For this, a needle injected into the participant s bone will remove marrow.
* Optional lymph node biopsy. For this, the participants whole lymph node or part of it will be removed through the skin.
* Optional lymphapheresis. For this, the participants blood is removed through a vein in one arm, the white blood cells separated out, and the blood returned through a vein in the other arm.

Participants will take duvelisib twice daily by mouth. They will continue ibrutinib at their current dose for the first 6 months. They will continue to take duvelisib until their CLL/SLL stops responding or they develop intolerable side effects.

Participants will take an antibiotic and antiviral medication. They may take steroids.

Participants will have blood tests every 2 weeks during the first 2 months.

Participants will have monthly follow-up visits during the first 6 months and every 3 months thereafter. These will include repeats of some of the screening tests.

DETAILED DESCRIPTION:
Background:

* In chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), ibrutinib resistance is predominantly caused by somatic mutations in BTK and PLCG2. Virtually all patients with detectable mutations eventually develop progressive disease. Patients who discontinue ibrutinib often have rapidly progressive disease that can be difficult to control. These observations suggest that BTK inhibitors still exert at least a partial anti-tumor effect. Outcomes after ibrutinib discontinuation are poor. Early detection of BTK and PLCG2 mutations represents an opportunity for preemptive intervention to eliminate the resistant clone.
* Duvelisib is a dual PI3K-gamma and delta inhibitor. Duvelisib monotherapy improved progression-free survival and overall response rate compared to ofatumumab and had a manageable safety profile in subjects with previously treated CLL/SLL. Based on these results, duvelisib received US approval for CLL/SLL after at least 2 prior therapies.
* This study will assess duvelisib in patients who develop disease progression or BTK and/or PLCG2 mutations on ibrutinib. Duvelisib will overlap with ibrutinib for the first six 28-day cycles to prevent disease acceleration often seen in patients who discontinue ibrutinib.

Primary Objective:

-To investigate the rate of overall response to duvelisib in patients with ibrutinib-resistant CLL.

Key Eligibility Criteria:

* Patients on current treatment for CLL/SLL with ibrutinib and at least one of the following:

  * BTK and/or PLCG2 mutations
  * Progressive CLL per CLL guidelines
* Patients with known Richter transformation will be excluded.

Design:

* This is a single-center, single-arm, open-label phase 2 study with a safety lead-in cohort.
* Treatment plan: Duvelisib will be administered with ibrutinib for the first six 28-day cycles then duvelisib monotherapy will be administered continuously until disease progression or intolerance.

Study Duration: 5 years.

Participant Duration: until disease progression or intolerance.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years
* Diagnosis of CLL or SLL as defined by the following:

  * CLL: clonal B cells greater than or equal to 5,000 cells/uL in the peripheral blood.
  * SLL: lymphadenopathy with histopathological evaluation consistent with SLL, absence of cytopenia caused by clonal marrow infiltrate, and <5,000 B cells/uL in the peripheral blood
  * Immunophenotype: co-expression of CD5, CD19, CD20, and CD23. CD23 negative cases may be included if there is an absence of t(11;14).
* Current treatment with ibrutinib for CLL.
* Mutations in BTK and/or PLCG2 (from a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory) with measurable disease characterized by at least 1 of the following:

  * Lymphadenopathy: greater than or equal to 1 lymph node measuring greater than or equal to 1.5 cm in the greatest diameter
  * Splenomegaly: spleen measuring > 13 cm in craniocaudal length
  * Lymphocytosis: greater than or equal to 5,000 B cells/ L
  * Bone marrow infiltration: CLL comprising greater than or equal to 30% of all cells

or

Progressive disease characterized by at least 1 of the following when compared with nadir values:

* Lymphadenopathy: appearance of any new enlarged lymph nodes (greater than or equal to 1.5 cm) or an increase by greater than or equal to 50% in greatest determined diameter of any previous site (greater than or equal to 1.5 cm).
* Splenomegaly: an increase in the cranio-caudal dimension of the spleen by greater than or equal to 2 cm from nadir, on imaging or physical exam.
* Lymphocytosis: an increase in the number of blood lymphocytes by greater than or equal to 50% over nadir with greater than or equal to 5,000 cells/uL B cells not attributable to redistribution of leukemia cells from lymphoid tissues to the blood related to treatment with kinase inhibitor.
* Cytopenia: occurrence of cytopenia directly attributable to CLL and unrelated to autoimmune cytopenia or treatment, as documented by a decrease of Hb levels greater than or equal to 2 g/dL or <10 g/dL, or by a decrease of platelet counts greater than or equal to 50% or <100,000/uL, if the marrow biopsy is consistent with the cytopenia resulting from increased marrow infiltration of clonal CLL cells.

  * Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
  * Adequate organ function as defined below

Hematological:

* Absolute neutrophil count (ANC) greater than or equal to 1000/uL
* Platelets greater than or equal to 75,000/uL

Renal:

-Serum creatinine < 2.0 mg/dL

Hepatic:

* Serum total bilirubin less than or equal to 1.5 X ULN except subjects with Gilbert's Syndrome
* AST (SGOT) and ALT (SGPT) less than or equal to 3.0 X ULN
* For women of childbearing potential (WCBP): negative serum beta human chorionic gonadotropin (beta-hCG) pregnancy test within 7 days before first treatment (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months for women >55 years of age)
* Willingness of male and female subjects who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of the study treatment and 3 months after the last dose of duvelisib
* Willingness and ability to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

EXCLUSION CRITERIA:

* Richter transformation of CLL into an aggressive lymphoma
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function
* Prior history of drug-induced colitis or pneumonitis
* Known hypersensitivity to any of the study drugs
* Major surgery within 4 weeks prior to screening
* Central nervous system (CNS) non-Hodgkin lymphoma (NHL); lumbar puncture not required unless CNS involvement is clinically suspected
* Active cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection (i.e., subjects with detectable viral load)
* Infection with hepatitis B or hepatitis C:

  * Subjects with a positive hepatitis B surface antigen (HBsAg)) will be excluded
  * Subjects with or hepatitis C antibody (HCV Ab) will be excluded, unless they have received curative treatment for hepatitis C virus (HCV) and have undetectable viral RNA by PCR.
  * Subjects with a positive hepatitis B core antibody (HBcAb) must have negative hepatitis B virus (HBV) deoxyribonucleic acid (DNA) to be eligible, must receive prophylaxis with entecavir (or equivalent) concomitant with duvelisib treatment, and must be periodically monitored for HBV reactivation by institutional guidelines
* Investigators who strongly believe that a positive HBcAb is false due to passive immunization from previous immunoglobulin infusion therapy should consider the risk-benefit for the patient given the potential for reactivation
* Infection with human immunodeficiency virus (HIV): Subjects must be receiving antiretroviral therapy, have undetectable HIV RNA viral load and CD4 cell count greater than or equal to 200/uL to be eligible, must continue antiretroviral therapy concomitant with duvelisib treatment, and must be periodically monitored for suppression of viral load and potential drug-drug interactions between antiretroviral therapy and duvelisib
* Infection with human T-lymphotropic virus type 1
* History of tuberculosis treatment within the 2 years prior to randomization
* History of chronic liver disease, veno-occlusive disease, alcohol abuse, or illicit drug use
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine) or systemic steroids >20 mg of prednisone (or equivalent) once daily (QD)
* Ongoing treatment for systemic bacterial, fungal, or viral infection at screening

NOTE: Subjects on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met

* Administration of a live or live attenuated vaccine within 6 weeks of randomization
* Concurrent administration of medications or foods that are strong inhibitors or inducers of cytochrome P450 3A (CYP3A). No prior use within 2 weeks before the start of study intervention.
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV) at screening
* Baseline left ventricular ejection fraction (LVEF) < 45 percent
* Baseline QT interval corrected with Fridericia's method (QTcF) > 500 ms

NOTE: criterion does not apply to subjects with a right or left bundle branch block (BBB)

* Subjects with clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea, vomiting, or any other condition that will interfere significantly with drug absorption
* Female subjects who are pregnant or breastfeeding
* Concurrent active malignancy that requires treatment except malignancies treated with antihormonal therapy alone, nonmelanoma skin cancer, or carcinoma in situ of the cervix.
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or a pacemaker within the last 6 months prior to screening
* Unstable or severe uncontrolled medical condition (e.g., unstable cardiac function, unstable pulmonary condition, uncontrolled diabetes and inflammatory GI diseases such as Crohn s Disease) or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the risk to the subject associated with his or her participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare C Sun, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-H-0016.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated prematurely due to unexpected sudden death on study.
Pre-assignment Details: Participants were enrolled on study based on safety lead-in with a 3+3 dose-escalation design.
Period: Overall Study
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Started | 3
Dose Level 1 | 3
Completed | 0
Not Completed | 3
Not completed — Death | 1
Not completed — Study Terminated Early | 2

BASELINE CHARACTERISTICS:
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Participant Overall Response Rate (ORR)
Description: Overall response rate with modification for treatment-related lymphocytosis. Response is defined below and followed iwCLL 2008 guidelines and incorporated clarifications for lymphocytosis associated with kinase inhibitors. Complete Response: Lymph Nodes = None greater or equal to 1.5 cm; Spleen &/or liver size = Spleen less than 13 cm &/or liver size normal; Blood Lymphocytes = less than 4000/μL. Partial Response: Lymph Nodes, Spleen and/or liver size, plus Blood Lymphocytes = Decrease greater than or equal to 50%. Partial Remission with Lymphocytosis: Lymph Nodes and Spleen and/or liver size = Decrease greater than or equal to 50%; Blood Lymphocytes = Increase or decrease greater than 50%. Progressive Disease: Lymph Nodes = Increase ≥ 50% or any new lesion > 1.5 cm; Spleen and/or liver size = Increase ≥ 50% or new splenomegaly; Blood Lymphocytes = Increase ≥ 50% and > 5000/μL B cells. Stable Disease: Lymph Nodes, Spleen and/or liver size plus Blood Lymphocytes =Change of -49% to +49%
Time Frame: After 12 weeks
Population: Intent-to-treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 3
Participants
  Complete Remission (CR) | 0
  Partial Remission (PR) | 0
  Partial Remission with lymphocytosis (PRL) | 0
  Progressive Disease (PD) | 0
  Stable Disease (SD) | 1

2. Secondary Outcome: Number of Participants With Progression-free Survival
Description: Number of participants with progression-free survival as defined as time from treatment initiation to progression of disease or death from any cause.
Time Frame: From Day 1 to progression of disease or death from any cause, which ever came first, assessed up to approximately 6 months
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 3
Participants
  Progression of Disease | 1
  Death | 1

3. Secondary Outcome: Participant Overall Survival
Description: Participant overall survival as defined as time from treatment initiation to death from any cause
Time Frame: From Day 1 to death from any cause, which ever came first, assessed up to approximately 6 months
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 3
Participants
  Death | 1
  Alive | 2

4. Secondary Outcome: Duration of Response in Days
Description: Duration of response in days as defined as time from initial response to progression of disease.
Time Frame: From initial response [12 weeks or later] to progression of disease
Population: Participants who have achieved response only
Groups:
- Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma: Duvelisib with ibrutinib will be administered for the first six 28-day (± 7) cycles followed by duvelisib alone until disease progression or intolerance. Duvelisib is an orally administered at 15 mg twice a day (dose level 1) or 25 mg twice day (dose level 2) or. Subjects will continue the same dose of ibrutinib prior to study enrollment for the first six 28-day cycles. Ibrutinib is an orally administered and provided as 140 mg white opaque capsules or tablets in 4 strengths: 140 mg, 280 mg, 420 mg, and 560 mg.
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Achieved Best Response
Description: Number of participants who achieved best response [complete response is better than partial response is better than stable disease].
  Complete Response: Lymph Nodes = None greater or equal to 1.5 cm; Spleen &/or liver size = Spleen less than 13 cm &/or liver size normal; Blood Lymphocytes = less than 4000/μL. Partial Response: Lymph Nodes, Spleen and/or liver size, plus Blood Lymphocytes = Decrease greater than or equal to 50%. Partial Remission with Lymphocytosis: Lymph Nodes and Spleen and/or liver size = Decrease greater than or equal to 50%; Blood Lymphocytes = Increase or decrease greater than 50%. Progressive Disease: Lymph Nodes = Increase ≥ 50% or any new lesion > 1.5 cm; Spleen and/or liver size = Increase ≥ 50% or new splenomegaly; Blood Lymphocytes = Increase ≥ 50% and > 5000/μL B cells. Stable Disease: Lymph Nodes, Spleen and/or liver size plus Blood Lymphocytes =Change of -49% to +49%
Time Frame: After greater than or equal to 3 cycles [12 weeks] of treatment, up to 6 months
Population: Participants who have had greater than or equal to one response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Safety of Duvelisib Plus Ibrutinib Combination and Duvelisib Monotherapy
Description: Safety as defined by number of dose limiting toxicities during first cycle of duvelisib plus ibrutinib combination and serious adverse events while participants are taking duvelisib plus ibrutinib combination followed by duvelisib monotherapy.
Time Frame: From time of informed consent to 30 days after last dose of duvelisib plus ibrutinib combination
Population: Intent-to-treat population
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 3
Number of Serious Adverse Events | 2

ADVERSE EVENTS:
Time Frame: 6 months
Description: All events whether volunteered by the patient, discovered by study personnel during questioning, or detected through physical examination, clinically significant laboratory test, or other means will be recorded in the patient's medical record.
Arm/Group | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (N=3)
Colitis (Gastrointestinal disorders) | 1 (1)
Sudden Death Not Otherwise Specified (NOS) (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duvelisib for Ibrutinib-Resistant Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04209621/Prot_SAP_002.pdf
  • Informed Consent Form (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04209621/ICF_000.pdf